CLINICAL TRIAL: NCT06318962
Title: Examining the Efficacy of a Digital Therapeutic to Prevent Suicidal Behaviors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UMemphis; SPC-1000007404 GR127268 (Other: Department of Defense)
Record Dates: First submitted 2024-02-26; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Suicidal Behaviors; Suicide Ideation; Depression/Anxiety
Keywords: BCBT; Suicide Ideation; Suicide Attempts; Depression and Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; Suicide, Attempted

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Therapeutic (Experimental): BCBT Delivery via digital app
  Interventions: Behavioral: Aviva
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: Aviva — Digital phone app for BCBT
  Arms: Digital Therapeutic

SUMMARY:
The primary aim of the project is to test the efficacy of BCBT delivered via a digital platform (i.e., smartphone) to Servicemembers with recent suicidal ideation and/or suicide attempts presenting to primary care clinics. Given existing challenges of scaling empirically-supported treatments/interventions for suicidality with fidelity, this project could lead to markedly expanded access to BCBT, along with improving our understanding about what intervention strategies are most effective and how they can be delivered with meaningful fidelity. Aviva, the digital version of BCBT, was developed for use with patients across the full spectrum of healthcare settings, including primary care. Aviva is not an emergency alert system, rather a digital platform for delivery of the full scope of BCBT treatment components. An open-label single group Phase I clinical trial has demonstrated the safety, tolerability, feasibility, fidelity, and potential efficacy of Aviva, with participants completing modules over 8 weeks, and follow-up assessments at weeks 1, 4, and 8. Subsequent refinements included the addition of technical features that would allow patients to revisit and/or repeat previously completed modules, along with integration of more characters for delivering video vignettes and greater opportunities for skills practice and treatment engagement. These modifications have further enhanced Aviva safety, tolerability, and fidelity, consistent with the original BCBT protocol. Not only is it hypothesized that Aviva will result in significantly larger reductions in severity of suicidal ideation than participants randomized to the control condition, but also that greater app engagement will be negatively correlated with severity of suicidal thinking. Moderators and mediators (i.e. suicidal beliefs, wish to live, impulsive decision-making) of intervention effects will also be examined. The study will be conducted at the primary care clinics at Fort Carson, with a goal of enrolling 720 patients across a two-year timeframe. Participants will be identified using each clinic's existing suicide risk assessment methods, including the PHQ-9 suicide risk item and a score of 1 or higher on the CSSRS Screener (Recent). Participants will be randomly assigned to one of two treatment conditions, Aviva or control (i.e., development of a safety plan consistent with local procedures and policies, along with referral for standard mental health care and suicide risk management in accordance with local policies and procedures). In an effort to address potential performance bias specific to smartphone use, participants in the control condition will download the Suicide Safety Plan app to their smartphones. Those in the Aviva condition will also complete weekly check-ins with Project 2 research clinicians to review treatment adherence, identify and respond to any logistical/operational problems, and respond to any unexpected emergencies and/or participant safety concerns. Participants will have up to five data points: baseline, 3, 6, 9, and 12 months. All data available from all participants and all time points will be included in the analyses, consistent with the intent-to-treat principle. Across our two previous clinical trials and our in-progress RCT, attrition during the first 12 months postbaseline was <30% and we anticipate similar rates in this trial.

DETAILED DESCRIPTION:
See Attached Documents

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* suicidal ideation within the past week and/or a suicide attempt within the past 30 days
* ability to complete the informed consent process
* ownership of either an Apple iPhone iOS 11 or higher or an Android smartphone OS 8.1 or higher

Exclusion Criteria:

* an inability to complete informed consent procedures (e.g., acute intoxication, altered consciousness)
* experiencing active psychosis or mania requiring hospitalization; (3) and inability to use a smartphone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Self Injurious Thoughts and Behaviors Interview Revised | At intake, 3 months, 6 months, 9 months and 12 months
  Suicide Attempts, self-injury and suicidal ideation

SECONDARY OUTCOMES:
Beck Scale for Suicide Ideation | At intake, 3 months, 6 months, 9 months and 12 months
  Suicidal ideation
Beck Hopelessness Scale | At intake, 3 months, 6 months, 9 months and 12 months
  Hopelessness

CONTACTS AND LOCATIONS:
Locations (1):
- Fort Carson, Colorado Springs, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bryan C.J., Rudd M.D. Guilford Press; 2018. Brief cognitive-behavioral therapy for suicide prevention.
- [Result] Rudd MD, Bryan CJ, Wertenberger EG, Peterson AL, Young-McCaughan S, Mintz J, Williams SR, Arne KA, Breitbach J, Delano K, Wilkinson E, Bruce TO. Brief cognitive-behavioral therapy effects on post-treatment suicide attempts in a military sample: results of a randomized clinical trial with 2-year follow-up. Am J Psychiatry. 2015 May;172(5):441-9. doi: 10.1176/appi.ajp.2014.14070843. Epub 2015 Feb 13. PMID 25677353
- [Result] Rojas SM, Gold SD, Bryan CJ, Pruitt LD, Felker BL, Reger MA. Brief Cognitive-Behavioral Therapy for Suicide Prevention (BCBT-SP) via Video Telehealth: A Case Example During the COVID-19 Outbreak. Cogn Behav Pract. 2022 May;29(2):446-453. doi: 10.1016/j.cbpra.2020.12.001. Epub 2021 Feb 4. PMID 34602808
- [Derived] Rudd MD, Wine M, Pedler R, Wright M, Gleason VL, Perez-Munoz A, Tuna B, Tempchin J, Flowers TA, Bryan CJ. Examining the efficacy of a digital therapeutic to prevent suicidal ideation and behaviors in a primary care setting: Design and methodology of a randomized controlled trial with military service members. Contemp Clin Trials. 2025 Nov;158:108107. doi: 10.1016/j.cct.2025.108107. Epub 2025 Oct 10. PMID 41076117